CLINICAL TRIAL: NCT00376454
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Tolerability of a 14 Day Treatment Course of GW493838 50mg Compared to Placebo in Subjects With Peripheral Neuropathic Pain
Brief Title: The Study of GW493838, an Adenosine A1 Agonist, in Peripheral Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1A20004
Record Dates: First submitted 2006-09-13; First posted 2006-09-14 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Neuropathic Pain
Keywords: neuropathic pain
MeSH Terms: conditions — Neuralgia

INTERVENTIONS:
Drug: GW493838

SUMMARY:
The purpose of this study was to determine the analgesic effect of GW493838 in patients with post-herpetic neuralgia or peripheral nerve injury caused by trauma or surgery.

ELIGIBILITY:
Inclusion criteria (subjects must meet all of the following criteria in order to be eligible for this study):

* Females of non-child-bearing potential
* diagnosis of peripheral neuropathic pain as a result of: postherpetic neuralgia (PHN) from shingles for at least 3 months duration OR focal neuropathic pain related to nerve injury caused by trauma or surgery
* defined area of pain

Exclusion criteria

* discontinue agents for the treatment of neuropathic pain
* unable to refrain from alcohol and sedative use during the study
* confounding chronic pain which could not be differentiated from the peripheral neuropathic pain under study
* intractable pain of unknown origin or active infection in the area of nerve injury.
* clinically significant medical history or abnormality found on physical examination, laboratory assessment or ECG at Screening or Baseline
* severe asthma that has required oral corticosteroid use in the last 12 months or the subject had severe asthma that required, at anytime, hospitalization or mechanical ventilation support.
* clinical evidence of major depression (by medical history) except those subjects controlled by SSRIs.
* a known allergy or hypersensitivity to any of the investigational products (including rescue analgesia- acetaminophen), or pharmacological class of the investigational product (i.e. adenosine) and/or investigational product excipients.
* a clinically significant abuse of substances, defined as: Patterns of substance intake consistent with disruption of normal function in society; Past or current impairment of organ function reasonably related to substance intake; Any indication of difficulty in abstaining from substances for the duration of the study.
* had previously participated in a clinical study during the past 30 days in which the subject was exposed to an investigational or non-investigational drug or device
* currently participating in another clinical study in which the subject was exposed to an investigational or non-investigational drug or device
* prior blood reduction (450 mL or more) during the previous 30 days
* at risk of non-compliance
* a woman of childbearing potential or a woman who was lactating.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113
Dates: Start 2002-11; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Pain intensity

SECONDARY OUTCOMES:
Safety Pain relief Global Impression of Change Pain quality Evoked pain intensity Area of allodynia Onset of effect Responder rate Rescue medication pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (31):
- United States (31):
  - GSK Clinical Trials Call Center, Huntsville, Alabama
  - GSK Clinical Trials Call Center, Hot Springs, Arizona
  - GSK Clinical Trials Call Center, Little Rock, Arkansas
  - GSK Clinical Trials Call Center, La Jolla, California
  - GSK Clinical Trials Call Center, Oceanside, California
  - GSK Clinical Trials Call Center, Boulder, Colorado
  - GSK Clinical Trials Call Center, Fort Lauderdale, Florida
  - GSK Clinical Trials Call Center, Fort Myers, Florida
  - GSK Clinical Trials Call Center, Palm Beach, Florida
  - GSK Clinical Trials Call Center, Palm Beach Gardens, Florida
  - GSK Clinical Trials Call Center, Pembroke Pines, Florida
  - GSK Clinical Trials Call Center, South Daytona, Florida
  - GSK Clinical Trials Call Center, St. Petersburg, Florida
  - GSK Clinical Trials Call Center, West Palm Beach, Florida
  - GSK Clinical Trials Call Center, Evansville, Indiana
  - GSK Clinical Trials Call Center, Lexington, Kentucky
  - GSK Clinical Trials Call Center, Louisville, Kentucky
  - GSK Clinical Trials Call Center, Covington, Louisiana
  - GSK Clinical Trials Call Center, Boston, Massachusetts
  - GSK Clinical Trials Call Center, Henderson, Nevada
  - GSK Clinical Trials Call Center, Lebanon, New Hampshire
  - GSK Clinical Trials Call Center, Ridgewood, New Jersey
  - GSK Clinical Trials Call Center, Albany, New York
  - GSK Clinical Trials Call Center, Asheville, North Carolina
  - GSK Clinical Trials Call Center, Winston-Salem, North Carolina
  - GSK Clinical Trials Call Center, Tulsa, Oklahoma
  - GSK Clinical Trials Call Center, Altoona, Pennsylvania
  - GSK Clinical Trials Call Center, Duncansville, Pennsylvania
  - GSK Clinical Trials Call Center, Richardson, Texas
  - GSK Clinical Trials Call Center, Tacoma, Washington
  - GSK Clinical Trials Call Center, Madison, Wisconsin